CLINICAL TRIAL: NCT00893334
Title: Evaluation of Limb-Girdle Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Collaborators: Carolinas Medical Center lead study site (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB#4463; MDA Grant: 129066
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Becker Muscular Dystrophy; Limb-Girdle Muscular Dystrophy, Type 2A (Calpain-3 Deficiency); Limb-Girdle Muscular Dystrophy, Type 2B (Miyoshi Myopathy, Dysferlin Deficiency); Limb-Girdle Muscular Dystrophy, Type 2I (FKRP-deficiency)
Keywords: Duchenne and Becker muscular dystrophy; muscular dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies, Limb-Girdle; Miyoshi myopathy; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected one time for DNA analysis.Only to confirm genotype if results are not available prior enrollement
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- BMD:: Patients diagnosed with Becker Muscular Dystrophy
- LGMD2A: patient diagnosed with Limb-Girdle Muscular Dystrophy, type 2A Calpain-3 deficiency
- LGMD2B: Patients diagnosed with Limb-Girdle Muscular Dystrophy, type 2B Miyoshi myopathy Dysferlin deficiency
- LGMD2I: Patients diagnosed with Limb-Girdle Muscular Dystrophy, type 2I FKRP-deficiency
- Control: Healthy Controls

SUMMARY:
The purpose of this study is to understand the biochemistry of different types of Limb-Girdle Muscular Dystrophy (LGMD) and to determine appropriate outcome measures for future clinical treatment trials for LGMD. It is being conducted at two sites in the Cooperative International Neuromuscular Research Group (CINRG). It involves a one day clinical evaluation at a participating institution that will take approximately four to six hours, and will involve strength testing and muscle functional testing by a physical therapist, an evaluation by a physician, pulmonary function testing, a complete cardiac evaluation with electrocardiogram (ECG or EKG) and echocardiogram (Echo), and involve two blood draws, one before the evaluation and one after the evaluation is complete. During the visit, the participant will be asked to fill out a couple of questionnaires asking questions about quality of life and activity limitations, as well as his/her understanding of their diagnosis with regards to etiology (or cause of their muscle disorder), genetics, and inheritance of their muscle disorder.

DETAILED DESCRIPTION:
Specific Aims:

Aim 1: Evaluate integrity of the extracellular matrix in patients with LGMD by measuring serum growth factors and cytokines and compare these to a disease control (BMD) and normal volunteers.

Aim 2: Measure growth factors and cytokines following medical evaluation and compare them to the baseline levels.

Aim 3: Discovery Aim for future multicenter clinical trials in LGMD. Aim 3A: Abstract medical records with particular emphasis on age of disease onset, initial clinical symptoms, progression and location of the muscular weakness, treatments attempted, and other medical complications. A review of the diagnostic testing performed will also be conducted.

Aim 3B: Perform complete clinical evaluation including anthropometric measures, evaluation of joint limitations, timed functional testing, muscle strength, pulmonary function, and a cardiac assessment.

Aim 3C: Determine patient understanding of diagnosis of LGMD and genetic testing results. A questionnaire will be generated that addresses the patient's understanding of his/her diagnosis as well as their understanding of genetic concepts of autosomal recessive inheritance, genes, molecular testing and implications for themselves as well as their family.

Aim 3D: Quality of Life (QOL) questionnaires will be administered. These will be used to identify functional limitations by the patients and compare those limitations with the clinical evaluation.

Study Description

Only one visit will be necessary for this study. The study visit includes:

1. Review of the informed consent form
2. Blood collection Blood will be collected for the following: DNA extraction to confirm genotype if not already performed; Muscle Enzymes before and after physical evaluation; and Growth factors and cytokines: before and after physical evaluation.
3. Medical history review
4. Physical Examination
5. Questionnaires: Participants will complete 3 questionnaires: Diagnosis and genetic testing, ACTIVLIM, and INQoL
6. Clinical Evaluator assessment which includes: Manual Muscle Testing, Quantitative Muscle Testing, Pulmonary Function Testing, Anthropometric measurements, and Timed and Functional testing
7. Cardiac evaluation will include: Electrocardiogram and Echocardiogram

Control subjects will be required to come to the test site to complete the informed consent process, clinical evaluator assessment, and have blood drawn before and after the clinical evaluator assessment. No other examinations or procedures will be performed on the control participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Diagnosis of LGMD2I, LGMD2A, LGMD2B, or BMD as determined by muscle biopsy immunohistochemistry, immunoblotting, or molecular analysis.
* Able to travel to study site
* Normal controls will be recruited as either friends of the study participants or through separate recruitment.

Exclusion Criteria:

* Unable to travel to study site.
* Do not have the diagnosis of LGMD2I, LGMD2A, LGMD2B, or BMD after review of clinical testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population will include all patients diagnosed LGMD2I, LGMD2A, LGMD2B, and BMD. BMD is an X-linked recessive condition that only affects males. It has been described in all ethnic backgrounds. LGMD2I, LGMD2A and LGMD2B are autosomal recessive conditions affecting both males and females of all ethnic backgrounds equally, both sexes and all ethnicities are expected to be equally represented. Clinical symptoms manifest in the second decade of life, therefore all participants will be over the age of 18. Healthy controls will be recruited to match the study population based on age, sex, and ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The measurement of growth factors (TGF-B, IGF-II) and cytokines (IL18, IL1A, and IL1B) between the different types of LGMD and BMD. | 12 months
The difference in the growth factors (TGF-B, IGF-II) and cytokines (IL18, IL1A, and IL1B) pre-evaluation and post-evaluation. | 12 months

SECONDARY OUTCOMES:
Evaluation of surrogate and clinically relevant outcome measures in LGMD. | 24 months
Quality of life questionnaires to correlate patient- perceived limitations in daily activities with the quantitative strength measurements and functional ability with timed testing. | 24 months
Evaluation of patient understanding in their diagnosis and genetic etiology of their diagnosis. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Tesi-Rocha, M.D., Principal Investigator — Cooperative International Neuromuscular Research Group; Susan Sparks, M.D., Ph.D., Principal Investigator — Levine Children's Hospital
Locations (2):
- United States (2):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Carolinas Medical Center, Charlotte, North Carolina

REFERENCES:
- See also: CINRG — http://www.cinrgresearch.org